CLINICAL TRIAL: NCT03175406
Title: Comparing the Accuracy of Manipal Cervical Scoring System and Modified Bishop Score in Predicting Successful Induction of Labor
Brief Title: Predicting the Outcomes of Labor Induction
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer of obstetrics and gynecology, Ain Shams University
Other Study IDs: ASU maternity hospital
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Manipal cervical scoring system
  Other Names: The Burnett modification of Bishop score

SUMMARY:
Pre induction assessment using bishop scoring system and Manipal cervical scoring system performed on 105 pregnant females

DETAILED DESCRIPTION:
preinduction cervical assessment using The Burnett modification of Bishop score with

1. Cervical dilatation in centimeters will be given a score of zero if dilatation less than 1cm, a score of 1 if 1-2 cm dilated, a score of 2 if more than 2 cm dilataion.
2. Length of the cervix will be given a score of zero if more than 2 cm, a score of 1 if 1-2 cm, a score of 2 if less than 1 cm.
3. Station of fetal head will be given a score of zero if -2 or higher , a score of 1 if -1, a score of 2 if zero or lower.
4. Consistency of the cervix will be given a score of zero if firm, a score of 1 if soft and a score of 2 if soft and stretchable.
5. Position of the cervix will be given a score of zero if posterior, a score of 1 if mid position and a score of 2 if anterior. So, a total score (sum of all scores) of zero at a minimum to 10 at a maximum can be estimated.

and also preinduction cervical assessment using transvaginal ultrasound and Manipal system where:

1. Length of the cervix will be given a score of zero if more than 3 cm, a score of 1 if 2-3 cm, a score of 2 if less than 2 cm.
2. Length of the funnel will be given a score of zero if absent, a score of 1 if ≤ 0.5 cm, a score of 2 if more than 0.5 cm.
3. width of the funnel will be given a score of zero if absent, a score of 1 if ≤ 0.5 cm, a score of 2 if more than 0.5 cm.
4. cervical position and shape will be given a score of zero if curved, a score of 2 if straight
5. Distance of presenting part to external os will be given a score of zero if more than 3 cm, a score of 1 if 2-3 cm, a score of 2 if less than 2 cm

ELIGIBILITY:
Inclusion Criteria:

1. Singleton gestation at 37 completed weeks or greater .
2. Cephalic presentation.
3. Longitudinal lie.
4. Living fetus.
5. Intact membrane

Exclusion Criteria:

1. Previous cesarean delivery or rupture uterus.
2. Antepartum hemorrhage including (abruptio placenta, placenta previa or vasa previa).
3. Abnormal fetal lie or presentation.
4. Pervious uterine surgery as myomectomy.
5. Category II, III non stress test.
6. Pelvic structural deformity.
7. Intrautrine growth retardation or macrosomia (estimated fetal weight ˃ than 4kg).
8. Patients who received any pre induction ripening.
9. Active genital herpes.
10. Invasive cervical carcinoma

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 105 females with singleton term pregnancy undergoing induction of labor
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
the occurrence of active labor | within one day of labor induction
  successful labor induction(IOL)

SECONDARY OUTCOMES:
The interval from onset of induction to active labor | 24 hours
  duration of induction
Successful vaginal delivery | 48 hours
The need for cesarean delivery (CS) | 24 hours
  indication of CS (fetal distress ,failed induction,...)
maternal and fetal complication associated with IOL | during induction ,labor, and 24 hours postpartum
  tachy systole, postpartum hemorrhage, fetal distress

CONTACTS AND LOCATIONS:
Overall Officials: Gasser M El-Bishry, MD,FRCOG, Study Chair — Professor; Ihab F Allam, MD, Study Director — Professor

IPD SHARING:
Plan to Share IPD: Undecided